**Desoximetasone 0.15% Topical Spray** 

Protocol / Study No. DSXS 1502 / 71542604

#### STATISTICAL ANALYSIS PLAN

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Maximal Use Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Atopic Dermatitis

Protocol Number: DSXS 1502 Novum Study Number: 71542604

### **Sponsor:**

Taro Pharmaceuticals U.S.A., Inc. 3 Skyline Drive, Hawthorne, NY 10532 USA

#### **Contract Research Organization:**

Novum Pharmaceutical Research Services 225 W. Station Square Drive, Suite 200 Pittsburgh, PA 15219

January 12, 2016

Final Version 1.0

Desoximetasone 0.15% Topical Spray

Protocol / Study No. DSXS 1502 / 71542604

## SAP FINAL VERSION APPROVALS

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Maximal Use Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Atopic Dermatitis

| Written By: | |
|---|---|
| Signature: Jianhua Liu, MSc Senior Biostatistician Novum Pharmaceutical Research Services | Date: 04/24/2017 |
| Reviewed By: Signature: Pina D'Angelo, MSc Senior Director, Scientific Affairs (Biostatistics) Novum Pharmaceutical Research Services | Date: 04/24/2017 |
| Approved By: Signature: | Date: 23 Apr 2017 |

**Desoximetasone 0.15% Topical Spray** 

Protocol / Study No. DSXS 1502 / 71542604

## **Revision History**

| VERSION | DATE | DESCRIPTION OF REVISIONS | REVISED BY |
|---|---|---|---|
| Draft 1.0 | May 10, 2016 | New Document | Jianhua Liu |
| Final 1.0 | January 12, 2017 | Incorporate client comments and finalize SAP | Jianhua Liu |

## **Desoximetasone 0.15% Topical Spray**

Protocol / Study No. DSXS 1502 / 71542604

#### **List of Abbreviations and Definition of Terms**

ADaM Analysis Data Model

AE Adverse Event
BP Blood Pressure
BSA Body Surface Area

C Celsius

CRF Case Report Form

CDISC Clinical Data Interchange Standards Consortium

CRO Contract Research Organization
EASI Eczema Area and Severity Index

F Fahrenheit

FDA Food and Drug Administration

HR Heart Rate Hg Mercury

HPA Hypothalamic Pituitary Adrenal

ICH International Conference on Harmonisation

IGA Investigator's Global Assessment

IND Investigational New Drug

LOCF Last Observation Carried Forward

MedDRA Medical Dictionary for Regulatory Activities

ITT Intent-to-Treat

LOCF Last Observation Carried Forward OGD The Office of Generic Drugs

PP Per-Protocol

SAE Serious Adverse Event
SAP Statistical Analysis Plan
SAS Statistical Analysis System
SDTM Study Data Tabulation Model
USA United States of America

**Desoximetasone 0.15% Topical Spray** 

Protocol / Study No. DSXS 1502 / 71542604

## **TABLE OF CONTENTS**

| 1. | INTRODUCTION | 7 |
|---|---|---|
| 2. | OBJECTIVES | 7 |
| 3. | OVERALL STUDY DESIGN | 7 |
| | RANDOMIZATION AND BLINDING | |
| 5. | SAMPLE SIZE | 10 |
| 6. | STUDY ENDPOINTS | 10 |
| 7. | STATISTICAL ANALYSIS METHODS | 11 |
| | 7.1 Baseline Characteristics | 11 |
| | 7.1.1 Subject Disposition | 11 |
| | 7.1.2 Demographic and Other Baseline Characteristics | 11 |
| | 7.1.3 Medical History | |
| | 7.1.4 Concomitant Medications | 12 |
| | 7.1.5 Pregnancy Test | 12 |
| | 7.2 Safety Analysis of Potential HPA Axis Suppression | 12 |
| | 7.3 Safety Analysis | 13 |
| | 7.3.1 Adverse Events | 13 |
| | 7.3.2 Vital Signs | 13 |
| | 7.3.3 Laboratory Evaluations | 14 |
| | 7.3.4 Investigator Global Assessment | 14 |
| | 7.3.5 Eczema Area and Severity Index Score (EASI) | 14 |
| | 7.3.6 Percent BSA Affected | 15 |
| | 7.3.7 Pruritus Assessment | 15 |
| | 7.4 Multiple Comparisons | 15 |
| | 7.5 Methods for Handling Missing Data | 15 |
| | 7.6 Interim Analyses | |
| 8. | TABLE, LISTING AND FIGURE SHELLS | 15 |
| | T16.1.9.1 Summary of Enrolled Patients | 17 |
| | T16.1.9.2 Summary of Protocol Deviations (Safety Population) | 18 |
| | T16.1.9.3 Summary of Patients Randomized, Included in Safety Analysis of Potential | |
| | HPA Axis Suppression by Study Center | |
| | T16.1.9.4 Summary of Demographic Data (Safety Population) | 20 |
| | T16.1.9.5 Summary of Frequency of HPA Axis Suppression at the End of Treatment | |
| | (Day 28) | 22 |
| | T16.1.9.5a Summary of Logistic Regression Analysis Results of HPA Axis | |
| | Suppression at the End of Treatment (Day 28) | 23 |
| | T16.1.9.6 Summary of Percent BSA Affected with Plaque Psoriasis (Safety | |
| | Population) | 24 |
| | T16.1.9.7 Summary of Frequency of Investigator Global Assessment (IGA) (Safety | |
| | Population) | 25 |
| | T16.1.9.8 Summary of Total Score - Eczema Area and Severity Index (EASI) (Safety | |
| | Population) | 26 |

| Desoximetasone 0.15% Topical Spray |
|------------------------------------|
|------------------------------------|

Protocol / Study No. DSXS 1502 / 71542604

| | T16.1.9.9 Overall Summary of Adverse Events (Safety Population) | 27 |
|---|---|---|
| | T16.1.9.10.1 Summary of Frequency of All Adverse Events by Body System (Safety | |
| | Population) | 28 |
| | T16.1.9.10.2 Summary of Frequency of All Adverse Events in $\geq$ 2% of Patients by | |
| | Body System (Safety Population) | 28 |
| | T16.1.9.11 Summary of Frequency of All Adverse Events by Severity (Safety | |
| | Population) | 29 |
| | T16.1.9.12 Summary of Frequency of All Adverse Events by Relationship (Safety | |
| | Population) | 30 |
| | T16.1.9.13 Summary of Frequency of Serious Adverse Events (Safety Population) | |
| | T16.1.9.14 Summary of Adverse Events by Treatment (Safety Population) | 32 |
| | T16.1.9.15 Summary of Shift Analysis of Clinical Laboratory Assessments | |
| | (Chemistry) from Baseline to Day 28 (Safety Population) | 33 |
| | T16.1.9.16 Summary of Shift Analysis of Clinical Laboratory Assessments | |
| | (Hematology) from Baseline to Day 28 (Safety Population) | 33 |
| | T16.1.9.17 Summary of Frequency of Pruritis Assessment (Safety Population) | |
| | L16.2.1 Listing of Discontinued Patients | 35 |
| | L16.2.2 Listing of Protocol Deviations. | 36 |
| | L16.2.3 Patients Excluded from Safety Analysis of Potential HPA Axis Suppression | 37 |
| | L16.2.4.1 Listing of Demographic Data | 38 |
| | L16.2.4.2 Listing of Medical History | 39 |
| | L16.2.4.3 Listing of Concomitant Medication. | 40 |
| | L16.2.5.1 Listing of Drug Administration | |
| | L16.2.5.2 Listing of Study Medication Weight | |
| | L16.2.6.1 Listing of Cortisol Response Test Results | |
| | L16.2.6.2 Listing of HPA Axis Suppression Follow-Up | |
| | L16.2.6.3 Listing of Investigator Global Assessment (IGA) | |
| | L16.2.6.4 Listing of Percent BSA Affected with Plaque Psoriasis | |
| | L16.2.6.5 Listing of Eczema Area and Severity Index (EASI) | |
| | L16.2.6.6 Listing of Pruritis Assessment | |
| | L16.2.7 Listing of Adverse Events by Cohort | |
| | L16.2.8.1 Listing of Positive Pregnancy Test Results | |
| | L16.2.8.2 Listing of Abnormal Vital Signs | 51 |
| | L16.2.8.3 Listing of Abnormal Physical Examination Results | |
| | L16.2.8.4 Listing of Clinical Hematology Laboratory Results | |
| | L16.2.8.5 Listing of Clinical Chemistry Laboratory Results | |
| 1( | ). APPENDICES | |
| | APPENDIX A: Body Surface Area Calculation | |
| | APPENDIX B: Eczema Area and Severity Index Score (EASI) | |
| | APPENDIX C: Investigator Global Assessment (IGA) | |
| | APPENDIX D: Cortisol Response Test | 60 |

**Desoximetasone 0.15% Topical Spray** 

Protocol / Study No. DSXS 1502 / 71542604

#### 1. INTRODUCTION

This Statistical Analysis Plan (SAP) is based on the final Clinical Study Protocol DSXS 1502 (Novum Study No. 71542604) Rev. 6 dated 09/06/2016. The SAP provides details on the planned statistical methodology for the analysis of the study data. The SAP also outlines the statistical programming specifications for the tables, listings and figures.

This SAP describes the study endpoints, derived variables, anticipated data transformations and manipulations, and other details of the analyses not provided in the study protocol. This SAP therefore outlines in detail all other aspects pertaining to the planned analyses and presentations for this study.

The following documents were reviewed in preparation of this SAP:

- Final Clinical Study Protocol DSXS 1502 (Novum Study No. 71542604) Rev. 6 dated 09/06/2016
- Case Report Form Version 1.0 for Novum Study No. 71542604 dated 10/07/2015

The reader of this SAP is encouraged to also read the clinical protocol for details on the conduct of this study, and the operational aspects of clinical assessments and timing for completing a patient in this study.

### 2. OBJECTIVES

- 1. The primary objective of this study is to evaluate the potential of desoximetasone 0.15% topical spray to suppress HPA axis function in patients with moderate to severe atopic dermatitis.
- 2. The secondary objectives are to evaluate the efficacy parameters and adverse event (AE) profile of desoximetasone 0.15% topical spray administered to patients with moderate to severe atopic dermatitis.

#### 3. OVERALL STUDY DESIGN

This open label, safety study is designed to evaluate the potential for adrenal suppression after maximal use treatment with desoximetasone 0.15% topical spray (Taro Pharmaceuticals, U.S.A.), for the treatment of moderate to severe atopic dermatitis.

Up to 70 eligible patients with atopic dermatitis that satisfy all eligibility criteria will be enrolled into the study at Visit 2. Patients must be overall in good health. They should have a current diagnosis of moderate to severe atopic dermatitis with IGA score of at least 3 or 4.

## **Desoximetasone 0.15% Topical Spray**

Protocol / Study No. DSXS 1502 / 71542604

Up to seventy (70) patients stratified by age with a confirmed diagnosis of moderate to severe atopic dermatitis with:

Cohort 1- 10-20 patients age 18 years and older with  $\geq 25\%$  body surface area (BSA) affected

Cohort 2- 10 -20 patients age 12-17 years of age with  $\geq$  25% body surface area (BSA) affected

Cohort 3- 5-1 0 patients age 6-11 years of age with  $\geq 35\%$  body surface area (BSA) affected

Cohort 4- 5-1 0 patients age 2-5 years of age with with  $\geq$  35% body surface area (BSA) affected

Cohort 5- 5-1 0 patients 6 months to 1 year of age with  $\geq$  35% body surface area (BSA) affected

Cohorts will be enrolled in sequential order. Each cohort will initiate enrollment once the previous cohort has reached the minimum number of patients and a safety analysis has been reviewed. Each cohort will be enrolled based on the availability of patients.

Each cohort will be reviewed for the potential of HPA axis suppression. If at least 50% of patients in each cohort experience HPA axis suppression once the minimum number of patients has been enrolled and completed the cohort, enrollment for that cohort will be stopped and no further cohorts will be initiated. If at least 35% of patients have experienced HPA axis suppression across cohorts combined during the study, enrollment will be discontinued and no other cohorts will be initiated. Cohort 2 will not begin until safety data has been reviewed for Cohort 1. The same process will be followed for each cohort until the study is complete.

Patients enrolled in the study will apply product twice a day, according to provided instructions, for a total of 28 days.

Patients will attend a total of 4 Clinic Visits as follows:

- Visit 1 (within 10 days prior to enrollment): Screening
- Visit 2 (Day 1): Enrollment
- Visit 3 (Day 14±2): Interim Visit
- Visit 4 (Day 28±2): End of Study or Early Termination

**Desoximetasone 0.15% Topical Spray** 

Protocol / Study No. DSXS 1502 / 71542604

**Figure 1 Study Schematic** 

| | Visit 1 | Visit 2 | Visit 3 | Visit 4 | Visit 5 |
|---|---|---|---|---|---|
| Day | (-10 to 0) | 1 | 14 ± 2 | 28 ± 2 | 42 ± 4 |
| Procedures | Screening (within 10 days before enrollment) Before 12 pm | Enrollment | Interim<br>Visit | End of<br>Study/Early<br>Termination<br>Before 12 pm | Telephone<br>Follow-Up<br>Visit |
| Informed Consent | X | | | | |
| Medical History and<br>Demographics | X | | | | |
| Vital Signs | X | X | X | X | |
| Pregnancy Test* | X | X | X | X | |
| Physical Exam | X | | | X | |
| % BSA Assessment | X | X | X | X | |
| IGA Score | X | X | X | X | |
| EASI Score | X | X | X | X | |
| Concomitant Medication | X | X | X | X | |
| Laboratory Evaluations | X | | | X | |
| Cortisol Response Test | X | | | X | |
| Confirm Inclusion/Exclusion<br>Criteria | X | X | | | |
| Dispense Sunscreen and<br>Wristband | | X | | | |
| Weigh and Dispense Study<br>Drug | | X | X | | |
| Collect and Weigh Study<br>Drug | | | X | X | |
| Dispense/Review Patient<br>Diary | | X | X | X | |
| Adverse Events | | | X | X | X |
| Evaluation of Patient<br>Compliance to the Protocol | | | X | X | |

<sup>\*</sup> Pregnancy test will be carried out for females of childbearing potential.

**Desoximetasone 0.15% Topical Spray** 

Protocol / Study No. DSXS 1502 / 71542604

#### 4. RANDOMIZATION AND BLINDING

Patients eligible for enrollment into the study will fall into one of five cohorts:

**Cohort 1-** 10-20 patients age 18 years and older with ≥ 25% body surface area (BSA) affected

Cohort 2- 10 -20 patients age 12-17 years of age with  $\geq 25\%$  body surface area (BSA) affected

Cohort 3- 5-1 0 patients age 6-11 years of age with  $\geq$  35% body surface area (BSA) affected

Cohort 4- 5-1 0 patients age 2-5 years of age with with  $\geq$  35% body surface area (BSA) affected

Cohort 5- 5-1 0 patients 6 months to 1 year of age with  $\geq 35\%$  body surface area (BSA) affected

At Visit 2 eligible patients will be enrolled to the study and assigned a patient number.

Cohorts will be enrolled in sequential order. Each cohort will initiate enrollment once the previous cohort has reached the minimum number of patients and a safety analysis has been reviewed. Each cohort will be enrolled based on the availability of patients.

Each cohort will be reviewed for the potential of HPA axis suppression. If at least 50% of patients in each cohort experience HPA axis suppression once the minimum number of patients has been enrolled and completed the cohort, enrollment for that cohort will be stopped and no further cohorts will be initiated. If at least 35% of patients have experienced HPA axis suppression across cohorts combined during the study, enrollment will be discontinued and no other cohorts will be initiated. Cohort 2 will not begin until safety data has been reviewed for Cohort 1. The same process will be followed for each cohort until the study is complete.

#### 5. SAMPLE SIZE

The sample size of 70 patients, stratified by age and % BSA, was based on recommendations of the FDA in IND 101789 Guidance Meeting that took place on 01/14/2015 and FDA Advice Letter dated 04/27/2015 (Reference 103740601).

#### 6. STUDY ENDPOINTS

## **Primary Outcome Measures:**

Hypothalamic Pituitary Adrenal (HPA) Axis Response to Cosyntropin demonstrating the absence or presence of adrenal suppression at the end of treatment.

**Desoximetasone 0.15% Topical Spray** 

Protocol / Study No. DSXS 1502 / 71542604

### **Secondary Outcome Measures:**

Hypothalamic Pituitary Adrenal (HPA) Axis Response to Cosyntropin demonstrating the presence of adrenal suppression at the end of treatment with %BSA as a covariate. %BSA will be assessed using instructions in Appendix A.

#### 7. STATISTICAL ANALYSIS METHODS

If not otherwise specified, statistical significance is defined as p<0.05 and is two-tailed. Data will be summarized with respect to demographic and baseline characteristics and safety variables.

For categorical variables, the number and percent of each category within a parameter will be calculated for non-missing data. For continuous variables, statistics will include n, mean, standard deviation, median, minimum and maximum values.

All statistical analyses will be conducted using SAS<sup>®</sup>, Version 9.4 or higher. Datasets will be prepared using headings from Clinical Data Interchange Consortium (CDISC) Study Data Tabulation Model (SDTM) implementation for human clinical trials and ADaM (Analysis Dataset Model).

#### 7.1 Baseline Characteristics

#### 7.1.1 Subject Disposition

The subject accountability and disposition information will be summarized by study cohort. The number of subjects enrolled, treated with study medication will be tabulated by study cohort. In addition, completion status and primary reason for withdrawal will be summarized by study cohort.

#### 7.1.2 Demographic and Other Baseline Characteristics

The cohorts will be compared for basic demographics (age, gender, ethnicity and race), baseline IGA, baseline EASI and baseline total BSA.

Summary tables by cohort will be presented. Continuous variables will be summarized using descriptive statistics (n, mean, standard deviation, median, minimum, maximum). Categorical variables will be summarized using frequencies and percentage.

Baseline comparability of the five cohorts will be presented using Chi-square test for the categorical variables, and Analysis of Variance for the continuous variables.

All data will be listed by cohort and patient.

**Desoximetasone 0.15% Topical Spray** 

Protocol / Study No. DSXS 1502 / 71542604

### 7.1.3 Medical History

At Visit 1, patients will be questioned about medical history, including acute and chronic medical history and medical history relevant to their atopic dermatitis, as well as all medication use within the past 12 weeks.

Medical history data will be listed by cohort and patient.

#### 7.1.4 Concomitant Medications

At Visits 1-4, patients will be questioned about current and concomitant medication over the past 12 weeks

All prior and concomitant medications taken since screening until the end of the study will be listed by cohort and patient.

## 7.1.5 Pregnancy Test

Urine pregnancy tests on women of child-bearing potential will be performed at Visits 1, 2, 3 and 4.

Positive pregnancy test results will be listed by cohort and patient.

### 7.2 Safety Analysis of Potential HPA Axis Suppression

Dosing will be twice a day for 28 days excluding the doses prior to the Cortisol Response Test (54 applications). All patients who are enrolled, use at least 42 doses of the study drug and have data from a post-treatment cortisol response test will be included in the analysis. Patients who have not used 42 doses of the study drug will be excluded from the primary analysis of HPA axis suppression.

The primary analysis of interest is the proportion of patients in each cohort who are considered to have demonstrated possible HPA axis suppression following treatment with the study medicationA logistic regression of the proportion of patients in the study with HPA axis suppression may be performed as exploratory analysis with % BSA affected as a covariate. This will depend on the distribution of the %BSA data collected. See Appendix D for results from the cortisol response test considered indicative of potential HPA axis suppression.

Cohorts will be enrolled in sequential order. Each cohort will initiate enrollment once the previous cohort has reached the minimum number of patients and a safety analysis has been reviewed. Each cohort will be enrolled based on the availability of patients.

Each cohort will be reviewed for the potential of HPA axis suppression. If at least 50% of patients in each cohort experience HPA axis suppression once the minimum number of patients

### **Desoximetasone 0.15% Topical Spray**

Protocol / Study No. DSXS 1502 / 71542604

has been enrolled and completed the cohort, enrollment for that cohort will be stopped and no further cohorts will be initiated. If at least 35% of patients have experienced HPA axis suppression across cohorts combined during the study, enrollment will be discontinued and no other cohorts will be initiated. Cohort 2 will not begin until safety data has been reviewed for Cohort 1. The same process will be followed for each cohort until the study is complete.

## 7.3 Safety Analysis

Safety analysis will be conducted on all patients who applied at least one dose of study drug.

#### 7.3.1 Adverse Events

All the adverse events (AEs) reported throughout the study will be coded and classified according to the MedDRA (Medical Dictionary for Regulatory Activities) coding dictionary (Version 17.0 or higher). Each adverse event is to be evaluated for date of start and end, seriousness, severity, causal relationship with the study drugs, action taken and outcome.

A summary table of the number and percent of patients with AEs by system organ class, preferred term, and cohort will be presented. Each patient will be counted only once within each preferred term.

A frequency summary table of the number of AEs by system organ class, preferred term, severity, and cohort will be presented. Severity will be classified as "Mild", "Moderate", or "Severe".

Similarly, a frequency summary table of the number of AEs by system organ class, preferred term, and relationship to a study drug, and cohort will be presented. Relationship to a study drug will be classified as "Not Related" or "Related" where "Related includes "Possible", "Probable", or "Definite".

Should sufficient data exist, adverse event frequencies will be compared between treatments using Fisher's exact test.

All AEs will be listed by cohort and patient.

#### 7.3.2 Vital Signs

The patient's vital signs will be recorded (heart rate, blood pressure, temperature and respiration rate) at Visit 1, 2, 3 and 4.

Abnormal vital signs will be listed by cohort and patient.

**Desoximetasone 0.15% Topical Spray** 

Protocol / Study No. DSXS 1502 / 71542604

### 7.3.3 Laboratory Evaluations

At Visit 1 and Visit 4 a blood sample will be collected for hematology and clinical chemistry testing. The testing panel should include as a minimum the following tests:

## Hematology

- Hematocrit
- White blood cell count
- Platelets
- Hemoglobin
- Red blood cell count
- Differential white cell count

#### Chemistry

- Alkaline phosphatase
- Total bilirubin
- Alanine transaminase
- Creatinine
- Aspartate transaminase
- Glucose
- Blood urea nitrogen

Shift analysis using the categories; below, above and within the laboratory normal range will be performed to identify any specific laboratory parameter that shows a trend toward potentially clinically significant changes.

All data will be listed by cohort and patient.

## 7.3.4 Investigator Global Assessment

At Visit 1 a visual inspection to confirm a diagnosis of chronic plaque psoriasis will be done. At each visit the Investigator will perform an Investigator Global Assessment (IGA). At Visit 1 the patient must have an IGA of 3 (moderate) or 4 (severe) for inclusion in the study.

Investigator Global Assessment will be summarized using frequency and percentage by cohort and visit.

Investigator Global Assessment will also be listed by cohort and patient.

## 7.3.5 Eczema Area and Severity Index Score (EASI)

Eczema Area and Severity Index Score will be assessed at each visit.

## **Desoximetasone 0.15% Topical Spray**

Protocol / Study No. DSXS 1502 / 71542604

EASI will be summarized using frequency and percentage by cohort and visit. EASI will also be listed by cohort and patient.

#### 7.3.6 Percent BSA Affected

The % BSA recorded at Visit 1, 2, 3 and 4 will be summarized descriptively by cohort and visit.

All data will be listed by cohort and patient.

#### 7.3.7 Pruritus Assessment

A frequency summary table comparing the severity of pruritus for each cohort will be presented by visit.

All data will be listed by cohort and patient.

#### 7.4 Multiple Comparisons

No multiple comparison adjustment will be made in this study.

## 7.5 Methods for Handling Missing Data

For demographic and baseline characteristics, each variable will be analyzed using all available data. Patients with missing data will be excluded only from analyses for which data are not available.

#### 7.6 Interim Analyses

There is no interim analysis planned in this study.

#### 8. TABLE, LISTING AND FIGURE SHELLS

The following shells are provided in order to provide a framework for the display of data from this study. These shells may not be reflective of every aspect of this study but are intended to show the general layout of the Tables, Listings and Figures that will be included in the final clinical study report. Tables, Listings and Figures are numbered following the ICH structure. Table headers, variables names and footnotes will be modified as needed following data analyses. All descriptive and inferential statistical analyses will be performed using SAS® statistical software Version 9.4 or higher, unless otherwise noted.

TABLE, LISTING AND FIGURE SHELLS

**T16.1.9.1 Summary of Enrolled Patients** 

| Patients | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Total |
|---|---|---|---|---|---|---|
| Screened | | | | | | XXX |
| Randomized | xxx | XXX | XXX | XXX | xxx | XXX |
| Completed Study | xxx | xxx | xxx | XXX | xxx | XXX |
| Terminated Early | XXX | XXX | XXX | XXX | XXX | XXX |
| Early Termination Reason | XXX | XXX | XXX | XXX | XXX | xxx |
| Adverse Event | XXX | XXX | XXX | XXX | XXX | XXX |
| Enrolled in error | XXX | XXX | XXX | XXX | XXX | XXX |
| Insufficient therapeutic response/treatment failure | XXX | xxx | xxx | XXX | XXX | XXX |
| Lost to follow-up | XXX | xxx | xxx | XXX | XXX | XXX |
| etc. | | | | | | |
| Other | xxx | xxx | xxx | XXX | xxx | xxx |

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542604\PDF\xxx

Created on: ddmmmyy hh:mm

T16.1.9.2 Summary of Protocol Deviations (Safety Population)

| | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 4 | Cohort 5 | Total |
|---|---|---|---|---|---|---|---|
| Total Patients with Protocol Deviations | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Total Deviations | xxx | xxx | xxx | xxx | xxx | xxx | xxx |
| Enrolled in Error | xxx | xxx | xxx | xxx | xxx | xxx | xxx |
| Lost to Follow-up | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Missed Visit | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Non-compliance with dosing requirements | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Outside Visit Window | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Restricted Medication Use | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| etc | | | | | | | |
| Other | xxx | xxx | xxx | xxx | xxx | xxx | XXX |

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542604\PDF\xxx

Created on: ddmmmyy hh:mm

T16.1.9.3 Summary of Patients Randomized, Included in Safety Analysis of Potential HPA Axis Suppression by Study Center

| Site | | • | | Total | • | Cohort 1 | Col | nort 2 | Coh | ort 3 | Co | hort 4 | Co | hort 5 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| No. | PI Name | Rando-<br>mized | Included | Rando-<br>mized | Included | Rando-<br>mized | Included | Rando-<br>mized | Included | Rando-<br>mized | Included | Rando-<br>mized | Included | |
| All | - | XX | xx(xx.x%) | XX | xx(xx.x%) | XX | xx(xx.x%) | XX | xx(xx.x%) | XX | xx(xx.x%) | XX | xx(xx.x%) | |
| xx<br>xx | xxxx<br>xxxx | xx<br>xx | xx (xx.x%)<br>xx(xx.x%) | xx<br>xx | xx(xx.x%)<br>xx(xx.x%) | XX<br>XX | xx(xx.x%)<br>xx(xx.x%) | XX<br>XX | xx(xx.x%)<br>xx(xx.x%) | xx<br>xx | xx(xx.x%)<br>xx(xx.x%) | XX<br>XX | xx(xx.x%)<br>xx(xx.x%) | |

Path: L:\Studies Sas Codes\Clinical Trial\71542604\PDF\xxx

Created on: ddmmmyy hh:mm

T16.1.9.4 Summary of Demographic Data (Safety Population)

| | | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total | |
|---|---|---|---|---|---|---|---|
| | | N=xx | N=xx | N=xx | N=xx | N=xx | P-value |
| Age (years) | n | XX | XX | XX | XX | XX | x.xxxx |
| | $Mean \pm SD$ | $xx.x \pm x.x$ | $xx.x \pm x.x$ | $xx.x \pm x.x$ | $xx.x \pm x.x$ | $xx.x \pm x.x$ | |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X | |
| | Range | xx-xx | XX-XX | XX-XX | xx-xx | XX-XX | |
| Age Groups | 2 - 11 | - | - | - | xx (100.0%) | - | |
| | 12 - 15 | - | - | xx (100.0%) | - | - | |
| | 16 - 17 | - | xx (xx.x%) | - | - | - | |
| | 18 - 19 | - | xx (xx.x%) | - | - | - | - |
| | 19 - 40 | xx (xx.x%) | - | - | - | - | |
| | 41 - 64 | xx (xx.x%) | - | - | - | - | |
| | 65 - 75 | xx (xx.x%) | - | - | - | - | |
| | > 75 | xx (xx.x%) | - | - | - | - | |
| Race | American Indian or Alaska Native | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | X.XXXX |
| | Asian | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | Black/African American | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | Native Hawaiian or other Pacific Islander | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | White | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | Other | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Ethnicity | Hispanic or Latino | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | X.XXXX |
| | Not Hispanic or Latino | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |

N= number of patients in the cohort; n= number of patient with data available; % is based on N

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542604\PDF\xxx

Created on: ddmmmyy hh:mm

T16.1.9.4 Summary of Demographic Data (Safety Population)

| | | Cohort 1<br>N=xx | Cohort 2<br>N=xx | Cohort 3 N=xx | Cohort 4<br>N=xx | Cohort 5<br>N=xx | Total<br>N=xx | P-value |
|---|---|---|---|---|---|---|---|---|
| Baseline Total BSA | n | xx | xx | xx | xx | xx | XX | X.XXXX |
| | $Mean \pm SD$ | $xx.x \pm x.x$ | $xx.x \pm x.x$ | $xx.x \pm x.x$ | $xx.x \pm x.x$ | $xx.x \pm x.x$ | $xx.x \pm x.x$ | |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | |
| | Range | xx-xx | xx-xx | xx-xx | xx-xx | xx-xx | xx-xx | |
| Baseline IGA | Clear | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | X.XXXX |
| | Almost Clear | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | Mild | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | Moderate | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| EASI | n | xx | xx | XX | XX | XX | XX | X.XXXX |
| | $Mean \pm SD$ | $xx.x \pm x.x$ | $xx.x \pm x.x$ | $xx.x \pm x.x$ | $xx.x \pm x.x$ | $xx.x \pm x.x$ | $xx.x \pm x.x$ | |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | |
| | Range | xx-xx | xx-xx | xx-xx | xx-xx | xx-xx | xx-xx | |

N= number of patients in the cohort; n= number of patient with data available; % is based on N

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542604\PDF\xxx

Created on: ddmmmyy hh:mm

T16.1.9.5 Summary of Frequency of HPA Axis Suppression at the End of Treatment (Day 28)

| HPA Axis<br>Suppression | All<br>N=xx | Cohort 1<br>N=xx | Cohort 2<br>N=xx | Cohort 3<br>N=xx | Cohort 4<br>N=xx | Cohort 5<br>N=xx |
|---|---|---|---|---|---|---|
| Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542604\PDF\xxx

Created on: ddmmmyy hh:mm

T16.1.9.5a Summary of Logistic Regression Analysis Results of HPA Axis Suppression at the End of Treatment (Day 28)

| | Odds Ratio | 95% Wald<br>Confidence Limits | Wald<br>Chi-Square | P-value |
|---|---|---|---|---|
| Cohort 1 vs. Cohort 2 | X.XXXX | x.xxxx, x.xxxx | X.XXXX | X.XXXX |
| Cohort 1 vs. Cohort 3 | X.XXXX | x.xxxx, x.xxxx | X.XXXX | x.xxxx |
| Cohort 1 vs. Cohort 4 | X.XXXX | x.xxxx, x.xxxx | X.XXXX | x.xxxx |
| Cohort 1 vs. Cohort 5 | x.xxxx | x.xxxx, x.xxxx | X.XXXX | x.xxxx |
| Cohort 2 vs. Cohort 3 | x.xxxx | x.xxxx, x.xxxx | X.XXXX | x.xxxx |
| Cohort 2 vs. Cohort 4 | x.xxxx | x.xxxx, x.xxxx | X.XXXX | x.xxxx |
| Cohort 2 vs. Cohort 5 | x.xxxx | x.xxxx, x.xxxx | X.XXXX | x.xxxx |
| Cohort 3 vs. Cohort 4 | x.xxxx | x.xxxx, x.xxxx | X.XXXX | x.xxxx |
| Cohort 3 vs. Cohort 5 | x.xxxx | x.xxxx, x.xxxx | x.xxxx | x.xxxx |
| Cohort 4 vs. Cohort 5 | x.xxxx | x.xxxx, x.xxxx | x.xxxx | x.xxxx |
| Baseline % BSA affected | x.xxxx | x.xxxx, x.xxxx | X.XXXX | x.xxxx |

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542604\PDF\xxx

Created on: ddmmmyy hh:mm

T16.1.9.6 Summary of Percent BSA Affected with Plaque Psoriasis (Safety Population)

| Visit | Statistic | $ \begin{array}{l} \text{Cohort 1} \\ (\mathbf{N} = \mathbf{x}\mathbf{x}) \end{array} $ | $ \begin{array}{c} \text{Cohort 2} \\ (\mathbf{N} = \mathbf{x}\mathbf{x}) \end{array} $ | Cohort 3 $(N = xx)$ | Cohort 4 $(N = xx)$ | Cohort 5 $(N = xx)$ |
|---|---|---|---|---|---|---|
| 1 | n | XX | XX | XX | XX | XX |
| | $Mean \pm SD$ | $xxx.x \pm xx.x$ | $xxx.x \pm xx.x$ | $xxx.x \pm xx.x$ | $xxx.x \pm xx.x$ | $xxx.x \pm xx.x$ |
| | Median | XXX.X | XXX.X | XXX.X | xxx.x | XXX.X |
| | Range | xxx - xxx | xxx - xxx | xxx - xxx | xxx - xxx | xxx - xxx |
| 2 | | | | | | |
| 3 | | | | | | |
| 4 | | | | | | |

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542604\PDF\xxx Created on: ddmmmyy hh:mm

T16.1.9.7 Summary of Frequency of Investigator Global Assessment (IGA) (Safety Population)

| Visit | Score | Cohort 1 $(N = xx)$ | $ \begin{array}{l} \text{Cohort 2} \\ (\mathbf{N} = \mathbf{x}\mathbf{x}) \end{array} $ | Cohort 3 $(N = xx)$ | Cohort 4 $(N = xx)$ | Cohort 5 $(N = xx)$ |
|---|---|---|---|---|---|---|
| 1 | 0 (Clear) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | 1 (Almost Clear) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | 2 (Mild Disease) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | 3 (Moderate<br>Disease) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | 4 (Severe Disease) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 2 | 0 (Clear) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | 1 (Almost Clear) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | 2 (Mild Disease) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | 3 (Moderate<br>Disease) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | 4 (Severe Disease) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

3

4

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542604\PDF\xxx Created on: ddmmmyy hh:mm

T16.1.9.8 Summary of Total Score - Eczema Area and Severity Index (EASI) (Safety Population)

| Visit | Statistic | $ \begin{array}{l} \text{Cohort 1} \\ (\mathbf{N} = \mathbf{x}\mathbf{x}) \end{array} $ | $ \begin{array}{c} \text{Cohort 2} \\ (\mathbf{N} = \mathbf{x}\mathbf{x}) \end{array} $ | Cohort 3 $(N = xx)$ | Cohort 4 $(N = xx)$ | Cohort 5 $(N = xx)$ |
|---|---|---|---|---|---|---|
| 1 | n | XX | XX | XX | XX | XX |
| | $Mean \pm SD$ | $xxx.x \pm xx.x$ | $xxx.x \pm xx.x$ | $xxx.x \pm xx.x$ | $xxx.x \pm xx.x$ | $xxx.x \pm xx.x$ |
| | Median | XXX.X | XXX.X | XXX.X | xxx.x | XXX.X |
| | Range | xxx - xxx | xxx - xxx | xxx - xxx | xxx - xxx | xxx - xxx |
| 2 | | | | | | |
| 3 | | | | | | |
| 4 | | | | | | |

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542604\PDF\xxx Created on: ddmmmyy hh:mm

T16.1.9.9 Overall Summary of Adverse Events (Safety Population)

| D | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Total |
|---|---|---|---|---|---|---|
| Description | N=xx | N=xx | N=xx | N=xx | N=xx | N=xx |
| Patients Randomized | XXX | XXX | XXX | XXX | XXX | XXX |
| Patients with at least one AE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Discontinued study drug due to above AE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| AEs reported | XXX | xxx | xxx | xxx | xxx | xxx |
| Mild | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Moderate | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Not Related | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Related | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Death | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Serious AE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Related = Possible, Probable, Definite

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542604\PDF\xxx

Created on: ddmmmyy hh:mm

T16.1.9.10.1 Summary of Frequency of All Adverse Events by Body System (Safety Population)

| <b>Body System</b> | MedDRA Term | Cohort | Events | Patients | Fisher's<br>p-value |
|---|---|---|---|---|---|
| Patients with at least one AE | Total | Cohort 1 (N=xx) | XX | xx (xx.x%) | x.xxxx |
| | | Cohort 2 (N=xx) | XX | xx (xx.x%) | |
| | | Cohort 3 (N=xx) | XX | xx (xx.x%) | |
| | | Cohort 4 (N=xx) | XX | xx (xx.x%) | |
| | | Cohort 5 (N=xx) | XX | xx (xx.x%) | |
| Ear and labyrinth disorders | Ear pain | Cohort 1 (N=xx) | XX | xx (xx.x%) | x.xxxx |
| | | Cohort 2 (N=xx) | XX | xx (xx.x%) | |
| | | Cohort 3 (N=xx) | XX | xx (xx.x%) | |
| | | Cohort 4 (N=xx) | XX | xx (xx.x%) | |
| | | Cohort 5 (N=xx) | XX | xx (xx.x%) | |

N = Total number of patient in each cohort; Percentage is based on total number of patients.

 $Path: L: \Studies\_Sas\_Codes \Clinical\ Trial \71542604 \PDF \end{tens} xx$ 

Created on: ddmmmyy hh:mm

T16.1.9.10.2 Summary of Frequency of All Adverse Events in ≥ 2% of Patients by Body System (Safety Population)

T16.1.9.11 Summary of Frequency of All Adverse Events by Severity (Safety Population)

| <b>Body System</b> | MedDRA Term | Cohort | Mild | Moderate | Severe |
|---|---|---|---|---|---|
| Patients with at least one AE | Total | Cohort 1 (N=xx) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | Cohort 2 (N=xx) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | Cohort 3 (N=xx) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | Cohort 4 (N=xx) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | Cohort 5 (N=xx) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Ear and labyrinth disorders | Ear pain | Cohort 1 (N=xx) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | Cohort 2 (N=xx) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | Cohort 3 (N=xx) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | Cohort 4 (N=xx) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | Cohort 5 (N=xx) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

N = Total number of events in each cohort; Percentage is based on total number of events.

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542604\PDF\xxx Created on: ddmmmyy hh:mm

T16.1.9.12 Summary of Frequency of All Adverse Events by Relationship (Safety Population)

| <b>Body System</b> | MedDRA Term | Cohort | Related | Not Related |
|---|---|---|---|---|
| Patients with at least one AE | Total | Cohort 1 (N=xx) | xx (xx.x%) | xx (xx.x%) |
| | | Cohort 2 (N=xx) | xx (xx.x%) | xx (xx.x%) |
| | | Cohort 3 (N=xx) | xx (xx.x%) | xx (xx.x%) |
| | | Cohort 4 (N=xx) | xx (xx.x%) | xx (xx.x%) |
| | | Cohort 5 (N=xx) | xx (xx.x%) | xx (xx.x%) |
| Ear and labyrinth disorders | Ear pain | Cohort 1 (N=xx) | xx (xx.x%) | xx (xx.x%) |
| | | Cohort 2 (N=xx) | xx (xx.x%) | xx (xx.x%) |
| | | Cohort 3 (N=xx) | xx (xx.x%) | xx (xx.x%) |
| | | Cohort 4 (N=xx) | xx (xx.x%) | xx (xx.x%) |
| | | Cohort 5 (N=xx) | xx (xx.x%) | xx (xx.x%) |

N = Total number of events in each cohort; Percentage is based on total number of events. Related = Possible, Probable, Definite

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542604\PDF\xxx Created on: ddmmmyy hh:mm

T16.1.9.13 Summary of Frequency of Serious Adverse Events (Safety Population)

| Body System | MedDRA | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 |
|---|---|---|---|---|---|---|
| | Term | N=xx | N=xx | N=xx | N=xx | N=xx |
| Injury, poisoning and procedural complications | Alcohol poisoning | XX | xx | xx | XX | xx |

 $Path: L: \Studies\_Sas\_Codes \Clinical\ Trial \71542604 \PDF \xxx$ 

Created on: ddmmmyy hh:mm

# T16.1.9.14 Summary of Adverse Events by Treatment (Safety Population)

#### Cohort 1

| | | Severity | | Relationship to Study Drug | |
|---|---|---|---|---|---|
| Body System<br>MedDRA Term | Mild<br>n (%) | Moderate<br>n (%) | Severe<br>n (%) | Related<br>n (%) | Not Related<br>n (%) |
| Total AEs (N=xxx) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Ear and labyrinth disorders<br>Ear pain | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) |
| Hypoacusis | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

N = Total AEs in Cohort 1; n (%) = Number of AEs (Percent of Total AEs in Cohort 1) Related = Possible, Probable, Definite

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542604\PDF\xxx Created on: ddmmmyy hh:mm

Page 1 of N

Programming Note: Similar tables will be created for other cohorts.

T16.1.9.15 Summary of Shift Analysis of Clinical Laboratory Assessments (Chemistry) from Baseline to Day 28 (Safety Population)

## Alanine Aminotransferase (U/L)

| | Cohort 1<br>(N=xx) | | | | Cohort 2<br>(N=xx) | | Cohort 3 Cohort 4 (N=xx) (N=xx) | | | ļ | Cohort 5<br>(N=xx) | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Baseline-><br>Endpoint | Low | Normal | High | Low | Normal | High | Low | Normal | High | Low | Normal | High | Low | Normal | High |
| Low | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) |
| Normal | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) |
| High | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) |

Table will continue for other lab parameters.

Similar table will be created for T16.1.9.18.

T16.1.9.16 Summary of Shift Analysis of Clinical Laboratory Assessments (Hematology) from Baseline to Day 28 (Safety Population)

T16.1.9.17 Summary of Frequency of Pruritis Assessment (Safety Population)

| Visit | Score | Cohort 1 $(N = xx)$ | Cohort 2 $(N = xx)$ | Cohort 3 $(N = xx)$ | Cohort 4 $(N = xx)$ | Cohort 5 $(N = xx)$ |
|---|---|---|---|---|---|---|
| 1 | None | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Mild | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Moderate | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 2 | None | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Mild | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Moderate | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

3

4

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542604\PDF\xxx Created on: ddmmmyy hh:mm

**L16.2.1 Listing of Discontinued Patients** 

| Cohort | Patient<br>Number | Discontinuation<br>Reason |
|---|---|---|
| Cohort 1 | XX-XXXX<br>XX-XXXX | Withdrawal by Subject<br>Lost to Follow-up |
| Cohort 2<br>Cohort 3<br>Cohort 4 | | |
| Cohort 5 | | |

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542604\PDF\xxx Created on: ddmmmyy hh:mm

**L16.2.2 Listing of Protocol Deviations** 

| Cohort | Patient<br>Number | <b>Event Description</b> |
|----------------------|-------------------|--------------------------------|
| Cohort 1 | xx-xxxx | Outside Visit Window (Visit 3) |
| Cohort 2 | | |
| Cohort 3<br>Cohort 4 | | |
| Cohort 5 | | |

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542604\PDF\xxx

Created on: ddmmmyy hh:mm
L16.2.3 Patients Excluded from Safety Analysis of Potential HPA Axis Suppression

| Cohort | Patient<br>Number | Exclusion Reason |
|---|---|---|
| Cohort 1 | xx-xxxx | Patient has not used 42 doses of the study drug |
| Cohort 2 | | |
| Cohort 3<br>Cohort 4<br>Cohort 5 | | |

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542604\PDF\xxx

Created on: ddmmmyy hh:mm

## L16.2.4.1 Listing of Demographic Data

| Cohort 1 xx-xxxx 30 Female Not Hispanic or Latino Black or African | |
|---|---|
| | American |
| Cohort 2 | |
| Cohort 3 | |
| Cohort 4 | |
| Cohort 5 | |

 $Path: L: \Studies\_Sas\_Codes \Clinical\ Trial \71542604 \PDF \xxx$ 

Created on: ddmmmyy hh:mm

# L16.2.4.2 Listing of Medical History

| Cohort | Patient<br>Number | System | Diagnosis or<br>Surgical<br>Procedure | Start Date | End Date | Ongoing |
|---|---|---|---|---|---|---|
| Cohort 1 | XX-XXXX | Gynecologic | Menopause | yyyy-mm-dd | yyyy-mm-dd | |

Cohort 2

Cohort 3

Cohort 4

Cohort 5

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542604\PDF\xxx

Created on: ddmmmyy hh:mm

# L16.2.4.3 Listing of Concomitant Medication

| Cohort | Patient<br>Number | Treatment<br>Area | Medication | Dosage | Frequency | Route | Start/End<br>Date | Indication |
|---|---|---|---|---|---|---|---|---|
| Cohort 1 | XX-XXXX | No | Lisinopril | 20 MG | QD | РО | yyyy-mm-dd /<br>yyyy-mm-dd | Hypertension |

Cohort 2

Cohort 3

Cohort 4

Cohort 5

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542604\PDF\xxx

Created on: ddmmmyy hh:mm

#### L16.2.5.1 Listing of Drug Administration

| | Patient | Date of | Date of | Total | Compliance |
|----------|---------|------------|------------|---------------|------------|
| Cohort | Number | First Dose | Last Dose | Doses Applied | (%) |
| Cohort 1 | XXXX | yyyy-mm-dd | yyyy-mm-dd | XX | XX.X |

Cohort 2

Cohort 3

Cohort 4

Cohort 5

#### Note to programmer:

Compliance = [Total number of applications] / [Planned number of applications] \* 100%, where Planned number of applications is determined as follows:

for subjects who completed the study successfully: 56 applications (28 days of twice daily dosing); for subjects who discontinued early: the minimum between 56 and [(Date of Discontinuation – Date of First Application)].

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542604\PDF\xxx Created on: ddmmmyy hh:mm

L16.2.5.2 Listing of Study Medication Weight

| | D-4'4 | Bott | de 1 | Bottle | Total | |
|---|---|---|---|---|---|---|
| Cohort | Patient<br>Number | Date<br>Dispensed | Weight<br>Dispensed<br>(g) | Date<br>Collected | Weight<br>Collected<br>(g) | Amount<br>Applied<br>(g) |
| Cohort 1 | XXXX | yyyy-mm-dd | XX | yyyy-mm-dd | XX | XXX |

Cohort 3

Cohort 4

Cohort 5

 $Path: L: \Studies\_Sas\_Codes \Clinical\ Trial \71542604 \PDF \xxx$ 

Created on: ddmmmyy hh:mm

# L16.2.6.1 Listing of Cortisol Response Test Results

## Cohort 1

| Patient<br>Number | Visit | Was a Cortisol<br>Response Test<br>conducted? | Date | Basal<br>Sample<br>Draw Time | Injection<br>Time | Post-<br>Injection<br>Draw<br>Time | Basal<br>Cortisol<br>Concentration<br>Level<br>(mcg/100ml) | Post Injection<br>Cortisol<br>Concentration<br>Level<br>(mcg/100ml) | | Have<br>HPA Axis<br>Suppression |
|---|---|---|---|---|---|---|---|---|---|---|
| XX-XXXX | 1 | Yes | yyyy-mm-dd | hh:mm | hh:mm | hh:mm | XXX | XXX | No | |
| | 4 | Yes | yyyy-mm-dd | hh:mm | hh:mm | hh:mm | XXX | XXX | | No |

Table will continue for other cohorts.

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542604\PDF\xxx

Created on: ddmmmyy hh:mm

# L16.2.6.2 Listing of HPA Axis Suppression Follow-Up

#### Cohort 1

| Patient<br>Number | Is The Patient Showing Signs<br>Or Symptoms Of HPA Axis<br>Suppression?/<br>Was a Cortisol Response<br>Test Conducted? | Follow-Up<br>Test | Date/<br>Basal Sample Draw Time/<br>Injection Time/<br>Post-Injection Draw Time | Basal<br>Cortisol<br>Concentration<br>Level<br>(mcg/100ml) | Post Injection<br>Cortisol<br>Concentration<br>Level<br>(mcg/100ml) | Still Show<br>Signs of<br>HPA Axis<br>Suppression? | Was the Patient Referred to an Endocrinologist |
|---|---|---|---|---|---|---|---|
| xx-xxxx | Yes/ Yes | Test 1 | yyyy-mm-dd / hh:mm /<br>hh:mm/ hh:mm | XXX | XXX | No | No |

Table will continue for other cohorts.

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542604\PDF\xxx

Created on: ddmmmyy hh:mm

# L16.2.6.3 Listing of Investigator Global Assessment (IGA)

| Cohort | Patient<br>Number | Visit 1 | Visit 2 | Visit 3 | Visit 4 / Early<br>Termination |
|---|---|---|---|---|---|
| Cohort 1 | xx-xxxx | 0 | 0 | 1 | 0 |
| Cohort 2<br>Cohort 3<br>Cohort 4<br>Cohort 5 | | | | | |

 $Path: L: \Studies\_Sas\_Codes \Clinical\ Trial \71542604 \PDF \xxx$ 

Created on: ddmmmyy hh:mm

# L16.2.6.4 Listing of Percent BSA Affected with Plaque Psoriasis

| Cohort | Patient<br>Number | Visit 1 | Visit 2 | Visit 3 | Visit 4 / Early<br>Termination | Baseline Total<br>BSA (m^2) |
|---|---|---|---|---|---|---|
| Cohort 1 | XX-XXXX | XXX | XXX | XXX | XXX | X.XX |

Cohort 2

Cohort 3

Cohort 4

Cohort 5

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542604\PDF\xxx

Created on: ddmmmyy hh:mm

L16.2.6.5 Listing of Eczema Area and Severity Index (EASI)

| Cohort | Patient<br>Number | Visit | Location | Erythema | Induration,<br>Papulation,<br>Edema | Lichenification | Excoriation | Total<br>Grade | Total<br>EASI<br>Score |
|---|---|---|---|---|---|---|---|---|---|
| Cohort 1 | xx-xxxx | 1 | Head/Neck | 0 | 0 | 0 | 0 | 0 | XXXX |
| | | | Upper Limbs | 0 | 0 | 0 | 0 | 0 | |
| | | | Trunk | 1 | 1 | 1 | 1 | 4 | |
| | | | Lower Limbs | 0 | 0 | 0 | 0 | 0 | |
| | | 2 3 | | | | | | | |
| Cohort 2<br>Cohort 3<br>Cohort 4<br>Cohort 5 | | 4 | | | | | | | |

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542604\PDF\xxx

Created on: ddmmmyy hh:mm

L16.2.6.6 Listing of Pruritis Assessment

| Cohort | Patient<br>Number | Visit 1 | Visit 2 | Visit 3 | Visit 4/Early<br>Termination |
|---|---|---|---|---|---|
| Cohort 1 | xx-xxxx | 0 (None) | 1 (Mild) | 1 (Mild) | 1 (Mild) |

Cohort 3

Cohort 4

Cohort 5

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542604\PDF\xxx Created on: ddmmmyy hh:mm

# L16.2.7 Listing of Adverse Events by Cohort

| Cohort | Patient<br>Number | Body System /<br>MedDRA Term /<br>AE Term | Treatmen<br>t Area | Start /End<br>Date | Severity | Relationship<br>to Study<br>Drug | Outcome | Action Taken/<br>Other Action<br>Taken | SAE? |
|---|---|---|---|---|---|---|---|---|---|
| Cohort 1 | XX-XXXX | Nervous system disorders / | No | yyyy-mm-dd / | Mild | Not Related | Recovered | Dose Not Changed/ | No |
| | | Headache / | | yyyy-mm-dd | | | | None | |
| | | Headache | | | | | | | |

Cohort 2

Cohort 3

Cohort 4

Cohort 5

Related = Possible, Probable, Definite

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542604\PDF\xxx

Created on: ddmmmyy hh:mm

L16.2.8.1 Listing of Positive Pregnancy Test Results

| Cohort | Patient<br>Number | Visit 1 | Visit 2 | Visit 3 | Visit 4 |
|----------|-------------------|----------|----------|----------|----------|
| Cohort 1 | xx-xxxx | Negative | Negative | Negative | Positive |

Cohort 3

Cohort 4

Cohort 5

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542604\PDF\xxx Created on: ddmmmyy hh:mm

L16.2.8.2 Listing of Abnormal Vital Signs

| Cohort | Patient<br>Number | Age | Visit | Vital Sign | Normal Range | Result |
|---|---|---|---|---|---|---|
| Cohort 1 | xx-xxxx | XXX | 1 | Diastolic BP | xxx - xxx | XXX |
| | | | 2<br>3<br>4 | | | |
| Cohort 2<br>Cohort 3<br>Cohort 4 | | | | | | |

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542604\PDF\xxx

Created on: ddmmmyy hh:mm

L16.2.8.3 Listing of Abnormal Physical Examination Results

| Cohort | Patient<br>Number | Visit | System | Results |
|----------|-------------------|-------|--------|-----------------|
| Cohort 1 | XX-XXXX | 1 | HEENT | Abnormal (Scar) |
| | | 2 | | |
| | | 3 | | |
| | | 4 | | |
| Cohort 2 | | | | |
| Cohort 3 | | | | |
| Cohort 4 | | | | |
| Cohort 5 | | | | |

 $Path: L: \Studies\_Sas\_Codes \Clinical\ Trial \71542604 \PDF \xxx$ 

Created on: ddmmmyy hh:mm

L16.2.8.4 Listing of Clinical Hematology Laboratory Results

| Cohort | Patient<br>Number | Visit | Hematocrit (unit) | WBC (unit) | Platelets (unit) | Hemoglobin (unit) | etc. |
|---|---|---|---|---|---|---|---|
| Cohort 1 | XX-XXXX | 1 | XXX | XXX | XXX | XXX | XXX |
| | | 4 | XXX | XXX | XXX | xxx (Low) | XXX |

Cohort 3

Cohort 4

Cohort 5

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542604\PDF\xxx Created on: ddmmmyy hh:mm

L16.2.8.5 Listing of Clinical Chemistry Laboratory Results

| Cohort | Patient<br>Number | Visit | Alkaline<br>Phosphatase<br>( <i>unit</i> ) | Alnine<br>Transaminase<br>(unit) | Aspartate<br>Transaminase<br>(unit) | Blood Urea<br>Nitrogen<br>( <i>unit</i> ) | etc. |
|---|---|---|---|---|---|---|---|
| Cohort 1 | XX-XXXX | 1 | XXX | XXX | xxx (High) | XXX | XXX |
| | | 4 | XXX | XXX | XXX | XXX | XXX |

Cohort 3

Cohort 4

Cohort 5

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542604\PDF\xxx Created on: ddmmmyy hh:mm

**Desoximetasone 0.15% Topical Spray** 

Protocol / Study No. DSXS 1502 / 71542604

#### 10. APPENDICES

#### **APPENDIX A: Body Surface Area Calculation**

#### **Total Body Surface Area Calculation**

To calculate the Total BSA the following procedure (Mosteller Formula<sup>13</sup>) should be followed.

Total Body Surface Area (BSA) in meters squared

$$m^2 = ((height (cm) x weight (kg)) / 3600)^{1/2}$$

It is preferable that the patient's height and weight be measured in cm and kg however if needed:

To convert inches (in) to centimeters (cm) the following conversion should be used

$$1 \text{ inch} = 2.54 \text{ cm}$$

To convert pounds (lbs) to kilograms (kg) the following conversion should be used

$$1 lb = 0.45 kg$$

The patient's height and weight should be reported to the nearest cm and nearest 0.5 kg. The BSA should be reported to the nearest second decimal place.

For example a patient who is 68 inches tall and weighs 180 lbs will have a reported BSA of:

#### **%BSA Affected**

To estimate the % BSA Affected, the Investigator should use the method of approximation:

The "Rule of Nines" provides a general estimation of total BSA for several anatomic areas (each arm = 9%, each leg = 18%, back = 18%, chest and abdomen = 18%, head =

## **Desoximetasone 0.15% Topical Spray**

Protocol / Study No. DSXS 1502 / 71542604

9%, groin = 1%). The Investigator may then visually estimate the proportion of the involved skin within each anatomic area and calculate the total percentage of BSA affected. In children, hips and legs are smaller and the head, neck and shoulders are larger, as a result, a modified "Rule of Nines" is used (see diagram below).

| Part | 1-4 year child<br>body<br>% of total | 5-9 year child<br>body<br>% of total | 10-14 year child<br>body<br>% of total | Adult body % of total |
|---|---|---|---|---|
| Arm | 9.5% | 9.5% | 9.5% | 9% |
| Head | 19% | 15% | 12% | 9% |
| Neck | 1770 | 1370 | 1% | 1% |
| Leg | 15% | 17% | 18% | 18% |
| Anterior trunk | 16% | 16% | 16% | 18% |
| Posterior trunk | 16% | 16% | 16% | 18% |



**Desoximetasone 0.15% Topical Spray** 

Protocol / Study No. DSXS 1502 / 71542604

#### APPENDIX B: Eczema Area and Severity Index Score (EASI)

The EASI is a composite score based on the severity of four different signs of atopic dermatitis in four different areas of the body multiplied by the percent of that specific body area affected multiplied by a weighting factor.

Erythema

0 = Clear No evidence of erythema 1 = Mild Definite light red coloration 2 = Moderate Moderate redness, but not dark

3 = Severe Dark red coloration

Induration/papulation/edema

0 = Clear No evidence of any induration/papulation/edema

1 = MildBarely perceptible elevation2 = ModerateClearly perceptible elevation3 = SevereMarked and extensive elevation

Lichenification

0 = Clear No evidence of lichenification

1 = Mild Slight thickening of skin discerible only by touch and with

skin markings minimally exaggerated

2 = Moderate Definite thickening of skin with skin marking exaggerated so

at they form a visible criss-cross or ridged pattern

3 = Severe Thickened skin with skin markings visibly portraying an

exaggerated criss-cross or ridged pattern

**Excoriation** 

0 = Clear No evidence of excoriation

1 = Mild Scant evidence of excoriation with no signs of deepers skin

damage (absence of erosion or crusts)

2 = Moderate Several linear marks of skin with some showing evidence of

deeper skin injury (erosion, crust visible)

3 = Severe Many erosive or crusty lesions present

The patient will be required to rate the severity of their pruritis (itching/scratching/discomfort) over the previous 24 hours using the following scale:

#### **Pruritis**

0 = None None

1 = Mild Occasional slight itching or scratching

2 = Moderate Constant or intermittent itching/scratching/discomfort which

is not disturbing sleep

#### **Desoximetasone 0.15% Topical Spray**

Protocol / Study No. DSXS 1502 / 71542604

3 = Severe

Bothersome itching/scratching/discomfort which is disturbing sleep

Eczema, induration, excoriation and lichenification are part of the EASI score but pruritis is not.

#### **EASI Score**

The EASI score is calculated as follows:

Head/neck  $(E + I + X + L) \times Area \times 0.1$  (in children ages 0-7, x 0.2)

Upper Limbs (E+I+X+L) x Area x 0.2 Trunk (E+I+X+L) x Area x 0.3

Lower Limbs  $(E + I + X + L) \times Area \times 0.4$  (in children ages 0-7, x 0.3)

EASI SCORE = SUM OF ABOVE 4 REGIONS

E: Erythema,

I: Induration/papulation/edema

X: Excoriation L: Lichenification

Severity is based on the Investigator's assessment of individual signs and symptoms 0 = none, 1 = mild, 2 = moderate, 3 = severe using the definitions above

The % of each body region affected is scored as the variable Area above in the EASI formula. For the 4 body regions (head/neck, upper limbs, trunk and lower limbs) if the:

```
Area = 0 if % affected is 0%

Area = 1 if % affected is 1 to 9%

Area = 2 if % affected is 10 to 29%

Area = 3 if % affected is 30 to 49%

Area = 4 if % affected is 50 to 69%

Area = 5 if % affected is 70 to 89%

Area = 6 if % affected is 90 to 100%
```

EASI Score can be presented to the nearest whole number (no decimals and all numbers should be rounded, 0.5 should be rounded up to the nearest whole number)

The minimum score would be 0 and the Maximum Score would be 72. To be eligible for participation in this study a patient must have an EASI of at least 15 at baseline.

**Desoximetasone 0.15% Topical Spray** 

Protocol / Study No. DSXS 1502 / 71542604

# **APPENDIX C: Investigator Global Assessment (IGA)**

To be eligible for inclusion in the study the IGA must be 3 or 4 at baseline. To be considered a Clinical Success the patient must score a 0, 1 at Visit 4.

| 0 | Clear | Minor, residual discoloration, no erythema or induration/papulation, no oozing/crusting |
|---|---|---|
| 1 | Almost Clear | Just perceptible erythema, with almost no induration/papulation and no oozing/crusting |
| 2 | Mild Disease | Definite pink erythema with mild induration/papulation and no oozing/crusting |
| 3 | Moderate<br>Disease | Red erythema with moderate induration/papulation and there may be some oozing/crusting |
| 4 | Severe<br>Disease | Dark/bright red erythema with severe induration/papulation with oozing/crusting |

**Desoximetasone 0.15% Topical Spray** 

Protocol / Study No. DSXS 1502 / 71542604

## **APPENDIX D: Cortisol Response Test**

This cortisol release test is modified from the procedure of Wood et al as described in the Product Label for Cortrosyn<sup>TM</sup> (cosyntropin) for injection (Amphstar Pharmaceuticals, Inc.).

The procedure is as follows:

- 1. A single 5 ml blood sample should be taken as the basal sample.
- 2. 0.25 mg (a single vial) of Cortrosyn<sup>TM</sup> (cosyntropin) should be reconstituted with 1.0ml of 0.9% sodium chloride injection USP injected intramuscularly. In patients under 3 years of age, 0.125mg of Cortrosyn<sup>TM</sup> will be used.
- 3. 30 minutes after the IM injection a second 5 ml blood sample should be obtained. The resulting two serum samples (at least 1 ml of serum in each) should be processed and labeled according to the instructions provided and sent the same day to ACM Global Laboratory for analysis of basal and post stimulated serum cortisol concentration.

At Visit 1 and Visit 4 all patients will have a cortisol response test performed. The resulting blood sample should be sent to ACM Global Laboratory for immediate testing.

#### Visit 1 Test

The results of the cortisol response test must be obtained prior to study drug being dispensed at Visit 2. Only patients with normal baseline (Visit 1) cortisol and adrenal function (see criteria below) should be enrolled in the study.

#### Visit 4 Test

The test at the End of Study visit should not be performed if the patient dosed within 12 hours.

A patient will be considered to have normal basal cortisol level and adrenal function if they meet all three criteria listed below under Normal. Failure to meet any of these criteria is indicative of abnormal adrenal function or potential HPA axis suppression.

| | Cortisol Results | |
|---|---|---|
| | Normal | Abnormal |
| Basal (pre Cortrosyn <sup>TM</sup> injection) | ≥ 5 mcg/100ml | < 5 mcg/100ml |
| 30 minutes post<br>Cortrosyn <sup>TM</sup> | $\geq$ basal value + 7 | < basal value + 7 |
| Cortrosyn <sup>TM</sup> injection | > 18 mcg/100ml | ≤ 18 mcg/100ml |

HPA Axis suppression will be defined as a 30 minute post Cortrosyn<sup>TM</sup> injection level cortisol level of  $\leq$  18 mcg/100ml. As the study treatment period will be over, any patients with results of

#### **Desoximetasone 0.15% Topical Spray**

Protocol / Study No. DSXS 1502 / 71542604

HPA axis suppression will be advised not to initiate any new steroid therapy, topical or otherwise, and to return to the site in 28 days at which time they will be assessed for HPA axis suppression.

Any patient presenting with symptoms of HPA axis suppression, such as nausea, headache, myalgia, fatigue or loose stool, will be referred to an endocrinologist. As an additional safety precaution, wristbands identifying the patient as someone suffering from adrenal suppression secondary to steroid withdrawal will be provided to alert medical personnel should any emergencies arise before adrenal function returns to normal.

If the results of the cortisol response test still show signs of HPA axis suppression 28 days after discontinuing therapy the patient will be asked to return in 28 days (56 days after discontinuing steroid therapy) for another follow-up test. If the patient is still showing signs of HPA axis suppression 56 days after discontinuing steroid therapy and presents with related symptoms, the patient will be referred to an endocrinologist.

If HPA axis suppression persists for 56 days after discontinuing steroid therapy, but the patient has no symptoms they will be asked to return in 28 days (84 days after discontinuing steroid therapy) for another follow-up test. If HPA axis suppression persists for 84 days after discontinuing steroid therapy patients will be referred to an endocrinologist regardless of symptoms.

Patients should not be subjected to Cortrosyn<sup>TM</sup> testing, or any other challenge to their adrenal response, any sooner than 4 weeks from their last Cortrosyn<sup>TM</sup> test.

Follow-Up Schedule for Patients showing signs of HPA Axis Suppression

| Days | HPA Results | Symptoms | Patient Course |
|-----------|-------------|-----------|-----------------------------|
| after d/c | | | |
| 28 | Normal | N/A | Study over |
| 28 | Abnormal | Yes | Refer to endocrinologist |
| 28 | Abnormal | No | Repeat test in 28 days |
| 56 | Normal | N/A | Study over |
| 56 | Abnormal | Yes | Refer to endocrinologist |
| 56 | Abnormal | No | Repeat test in 28 days |
| 84 | Normal | N/A | Study over |
| 84 | Abnormal | Yes or No | Refer to an endocrinologist |